CLINICAL TRIAL: NCT00883129
Title: Mycophenolate vs. Oral Cyclophosphamide in Scleroderma Interstitial Lung Disease (Scleroderma Lung Study II)
Brief Title: Comparison of Therapeutic Regimens for Scleroderma Interstitial Lung Disease (The Scleroderma Lung Study II)
Acronym: SLSII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Roth (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Michael Roth, Professor, Division of Pulmonary & Critical Care; Vice Chairman for Research Compliance, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 632; R01HL089901 (NIH); R01HL089758 (NIH)
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Scleroderma; Interstitial Lung Disease
Keywords: Systemic Sclerosis; Mycophenolate Mofetil; Cyclophosphamide; High Resolution Computerized Tomography; Pulmonary Function; Dyspnea; Health Related Quality of Life
MeSH Terms: conditions — Scleroderma, Diffuse; Lung Diseases, Interstitial; Scleroderma, Systemic; Dyspnea | interventions — Mycophenolic Acid; Cyclophosphamide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Arm (Experimental): Participants will receive oral mycophenolate mofetil for 2 years.
  Interventions: Drug: Mycophenolate mofetil
- Cyclophosphamide Arm (Experimental): Participants will receive oral cyclophosphamide for 1 year, followed by placebo for 1 year.
  Interventions: Drug: Cyclophosphamide; Drug: Placebo

INTERVENTIONS:
Drug: Mycophenolate mofetil — 24 months of oral mycophenolate mofetil, up to a maximal dose of 1.5 grams twice daily as tolerated
  Other Names: CellCept
  Arms: Mycophenolate Arm
Drug: Cyclophosphamide — 12 months of oral cyclophosphamide, up to a maximal dose of 2 mg/kg daily as tolerated
  Other Names: Cytoxan
  Arms: Cyclophosphamide Arm
Drug: Placebo — 12 months of placebo will be delivered to participants in the Cyclophosphamide arm during the second year in order to maintain the blind with the Mycophenolate arm, which receives drug for the entire 2 years.
  Other Names: Sugar Pill
  Arms: Cyclophosphamide Arm

SUMMARY:
Scleroderma is a rare, long-term autoimmune disease in which normal tissue is replaced with dense, thick fibrous tissue. Normally, the immune system helps defend the body against disease and infection. In people with scleroderma, the immune system triggers fibroblast cells to produce too much of the protein collagen. The extra collagen becomes deposited in the skin and organs, causing hardening and thickening that is similar to the scarring process. Although scleroderma most often affects the skin, it also can affect other parts of the body, including the lungs, and in its most severe forms scleroderma can be life-threatening. Scleroderma-related interstitial lung disease is one example of a life-threatening scleroderma condition. In people with symptomatic scleroderma-related interstitial lung disease, scarring occurs in the delicate lung tissue, compromising lung function. The purpose of this study is to determine whether people with symptomatic scleroderma-related interstitial lung disease experience more respiratory benefits from treatment with a 2-year course of mycophenolate mofetil or treatment with a 1-year course of oral cyclophosphamide.

DETAILED DESCRIPTION:
Interstitial lung disease describes a condition in which the lung tissue has become scarred or inflamed. Interstitial lung disease caused by scleroderma, specifically seen as progressive pulmonary fibrosis, occurs in approximately 40 percent of patients with scleroderma and has emerged as the leading overall cause of death.

In a previous study, the Scleroderma Lung Study I (SLS I), investigators evaluated a 1-year cyclophosphamide (CYC) treatment for people with scleroderma-related interstitial lung disease. The study results demonstrated statistically significant improvements in forced vital capacity, total lung capacity, dyspnea, Rodnan skin scores, and several measures of quality of life. However, when patients were followed for another year after completing their CYC therapy, the beneficial effects of CYC waned and were no longer significant by the 24-month follow-up. Preliminary information suggests that an alternative immunosuppressive medication, mycophenolate mofetil (MMF), may be effective in treating this disease, be given for longer periods, and result in fewer side effects.

This study, the Scleroderma Lung Study II (SLS II), will compare the safety and efficacy of a 2-year treatment with MMF versus a 1-year treatment with CYC. Specifically, investigators will determine whether MMF produces similar or better improvements in lung capacity and fewer side effects throughout the entire 2-year period.

Participation will include about 21 study visits over a 2-year period. Eligible participants will be randomly assigned to receive either MMF twice daily for 2 years or CYC once daily for 1 year, followed by placebo for 1 year. Blood and urine samples will be collected every 2 weeks for the first 2 months and then once a month for the remainder of the study. Every 3 months, participants will attend study visits that will include pulmonary function tests, blood and urine sampling, a physical exam, and questionnaires about current health and medications. At the final study visit, participants will also undergo a high resolution computerized tomography (HRCT) scan and possibly a punch biopsy.

ELIGIBILITY:
Inclusion Criteria:

* The presence of either limited (cutaneous thickening distal but not proximal to elbows and knees, with or without facial involvement) or diffuse (cutaneous thickening proximal to elbows and knees, often involving the chest or abdomen) scleroderma, as determined by American College of Rheumatology criteria
* Dyspnea on exertion (grade 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index)
* FVC less than or equal to 80 percent of predicted value at screening and less than or equal to 85 percent predicted at baseline
* Onset of the first non-Raynaud manifestation of SSc within the prior 84 months
* Presence of any ground glass opacification on thoracic high resolution computerized tomography (HRCT)
* Repeat FVC at the baseline visit (Visit 2) within 10 percent of the FVC measured at screening and less than or equal to 85 percent predicted.

Exclusion Criteria:

* FVC less than 45 percent of predicted value at either screening or baseline
* Carbon monoxide diffusing capacity (DLCO) (HBg-corrected) less than 30 percent of predicted value and less than 40 percent of predicted when documentation of pulmonary artery pressures by echocardiogram, right heart catheterization or magnetic resonance imaging identifies clinically significant pulmonary hypertension. All participants with a DLCO less than 40 percent predicted must have documentation of pulmonary artery pressures in order to be considered for inclusion.
* FEV1/FVC ratio less than 65 percent at either screening or baseline
* Clinically significant abnormalities on HRCT not attributable to scleroderma
* Diagnosis of clinically significant resting pulmonary hypertension requiring treatment, as ascertained before study evaluation or as part of a standard of care clinical assessment performed outside of the study protocol
* Persistent unexplained hematuria (more than 10 red blood cells per high-power field [RBCs/hpf])
* History of persistent leukopenia (white blood cell count less than 4000) or thrombocytopenia (platelet count less than 150,000)
* Clinically significant anemia (less than 10g/dl)
* Baseline liver function test (LFTs) or bilirubin more than 1.5 times the upper limit of normal, other than that due to Gilbert's disease
* Concomitant and present use of captopril
* Serum creatinine more than 2.0mg/dL
* Uncontrolled congestive heart failure
* Pregnancy (documented by urine pregnancy test) and/or breast feeding
* Prior use of oral CYC or MMF for more than 8 weeks or the receipt of more than two intravenous doses of CYC in the past
* Use of CYC and/or MMF in the 30 days before random assignment
* Active infection (lung or elsewhere) whose management would be compromised by CYC or MMF
* Other serious concomitant medical illness (e.g., cancer), chronic debilitating illness (other than scleroderma), or unreliability or drug abuse that might compromise the patient's participation in the study
* Current use, or use within the 30 days prior to random assignment, of prednisone (or equivalent) in doses of more than 10 mg/day
* If of child bearing potential (a female participant <55 years of age who has not been postmenopausal for > 5 years and who has not had a hysterectomy and/or oophorectomy), failure to employ two reliable means of contraception (which may include surgical sterilization, barrier methods, spermicidals, intrauterine devices, and/or hormonal contraception).
* Use of contraindicated medications; more information on this criterion can be found in the study protocol
* Smoking of cigars, pipes, or cigarettes in the 6 months before study entry
* Use of medications with putative disease-modifying properties within the past month (e.g., D-penicillamine, azathioprine, methotrexate, Potaba)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald P. Tashkin, MD, Principal Investigator — University of California, Los Angeles; Robert M. Elashoff, PhD, Principal Investigator — UCLA School of Public Health; Michael D. Roth, MD, Principal Investigator — University of California, Los Angeles
Locations (14):
- United States (14):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Feinberg School of Medicine, Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, College of Medicine, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Medicine and Dentistry of New Jersey, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Medical School at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Li G, Gjertson D, Elashoff R, Shah SK, Ochs R, Vasunilashorn F, Abtin F, Brown MS, Goldin JG. Classification of parenchymal abnormality in scleroderma lung using a novel approach to denoise images collected via a multicenter study. Acad Radiol. 2008 Aug;15(8):1004-16. doi: 10.1016/j.acra.2008.03.011. PMID 18620121
- [Background] Elashoff RM, Li G, Li N. An approach to joint analysis of longitudinal measurements and competing risks failure time data. Stat Med. 2007 Jun 30;26(14):2813-35. doi: 10.1002/sim.2749. PMID 17124698
- [Background] Elashoff RM, Li G, Li N. A joint model for longitudinal measurements and survival data in the presence of multiple failure types. Biometrics. 2008 Sep;64(3):762-771. doi: 10.1111/j.1541-0420.2007.00952.x. Epub 2007 Dec 20. PMID 18162112
- [Background] Li N, Elashoff RM, Li G. Robust joint modeling of longitudinal measurements and competing risks failure time data. Biom J. 2009 Feb;51(1):19-30. doi: 10.1002/bimj.200810491. PMID 19197956
- [Background] Hant FN, Ludwicka-Bradley A, Wang HJ, Li N, Elashoff R, Tashkin DP, Silver RM; Scleroderma Lung Study Research Group. Surfactant protein D and KL-6 as serum biomarkers of interstitial lung disease in patients with scleroderma. J Rheumatol. 2009 Apr;36(4):773-80. doi: 10.3899/jrheum.080633. Epub 2009 Mar 13. PMID 19286849
- [Background] Kim HG, Tashkin DP, Clements PJ, Li G, Brown MS, Elashoff R, Gjertson DW, Abtin F, Lynch DA, Strollo DC, Goldin JG. A computer-aided diagnosis system for quantitative scoring of extent of lung fibrosis in scleroderma patients. Clin Exp Rheumatol. 2010 Sep-Oct;28(5 Suppl 62):S26-35. Epub 2010 Nov 3. PMID 21050542
- [Background] Furst DE, Tseng CH, Clements PJ, Strange C, Tashkin DP, Roth MD, Khanna D, Li N, Elashoff R, Schraufnagel DE; Scleroderma Lung Study. Adverse events during the Scleroderma Lung Study. Am J Med. 2011 May;124(5):459-67. doi: 10.1016/j.amjmed.2010.12.009. PMID 21531236
- [Background] Roth MD, Tseng CH, Clements PJ, Furst DE, Tashkin DP, Goldin JG, Khanna D, Kleerup EC, Li N, Elashoff D, Elashoff RM; Scleroderma Lung Study Research Group. Predicting treatment outcomes and responder subsets in scleroderma-related interstitial lung disease. Arthritis Rheum. 2011 Sep;63(9):2797-808. doi: 10.1002/art.30438. PMID 21547897
- [Background] Khanna D, Tseng CH, Farmani N, Steen V, Furst DE, Clements PJ, Roth MD, Goldin J, Elashoff R, Seibold JR, Saggar R, Tashkin DP. Clinical course of lung physiology in patients with scleroderma and interstitial lung disease: analysis of the Scleroderma Lung Study Placebo Group. Arthritis Rheum. 2011 Oct;63(10):3078-85. doi: 10.1002/art.30467. PMID 21618205
- [Background] Kim HJ, Brown MS, Elashoff R, Li G, Gjertson DW, Lynch DA, Strollo DC, Kleerup E, Chong D, Shah SK, Ahmad S, Abtin F, Tashkin DP, Goldin JG. Quantitative texture-based assessment of one-year changes in fibrotic reticular patterns on HRCT in scleroderma lung disease treated with oral cyclophosphamide. Eur Radiol. 2011 Dec;21(12):2455-65. doi: 10.1007/s00330-011-2223-2. Epub 2011 Sep 17. PMID 21927793
- [Background] Theodore AC, Tseng CH, Li N, Elashoff RM, Tashkin DP. Correlation of cough with disease activity and treatment with cyclophosphamide in scleroderma interstitial lung disease: findings from the Scleroderma Lung Study. Chest. 2012 Sep;142(3):614-621. doi: 10.1378/chest.11-0801. PMID 22156609
- [Result] Tashkin DP, Elashoff R, Clements PJ, Goldin J, Roth MD, Furst DE, Arriola E, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M; Scleroderma Lung Study Research Group. Cyclophosphamide versus placebo in scleroderma lung disease. N Engl J Med. 2006 Jun 22;354(25):2655-66. doi: 10.1056/NEJMoa055120. PMID 16790698
- [Result] Khanna D, Clements PJ, Furst DE, Chon Y, Elashoff R, Roth MD, Sterz MG, Chung J, FitzGerald JD, Seibold JR, Varga J, Theodore A, Wigley FM, Silver RM, Steen VD, Mayes MD, Connolly MK, Fessler BJ, Rothfield NF, Mubarak K, Molitor J, Tashkin DP; Scleroderma Lung Study Group. Correlation of the degree of dyspnea with health-related quality of life, functional abilities, and diffusing capacity for carbon monoxide in patients with systemic sclerosis and active alveolitis: results from the Scleroderma Lung Study. Arthritis Rheum. 2005 Feb;52(2):592-600. doi: 10.1002/art.20787. PMID 15692967
- [Result] Khanna D, Yan X, Tashkin DP, Furst DE, Elashoff R, Roth MD, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M, Clements PJ; Scleroderma Lung Study Group. Impact of oral cyclophosphamide on health-related quality of life in patients with active scleroderma lung disease: results from the scleroderma lung study. Arthritis Rheum. 2007 May;56(5):1676-84. doi: 10.1002/art.22580. PMID 17469162
- [Result] Clements PJ, Roth MD, Elashoff R, Tashkin DP, Goldin J, Silver RM, Sterz M, Seibold JR, Schraufnagel D, Simms RW, Bolster M, Wise RA, Steen V, Mayes MD, Connelly K, Metersky M, Furst DE; Scleroderma Lung Study Group. Scleroderma lung study (SLS): differences in the presentation and course of patients with limited versus diffuse systemic sclerosis. Ann Rheum Dis. 2007 Dec;66(12):1641-7. doi: 10.1136/ard.2007.069518. Epub 2007 May 7. PMID 17485423
- [Result] Tashkin DP, Elashoff R, Clements PJ, Roth MD, Furst DE, Silver RM, Goldin J, Arriola E, Strange C, Bolster MB, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel D, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M, Khanna D, Li N, Li G; Scleroderma Lung Study Research Group. Effects of 1-year treatment with cyclophosphamide on outcomes at 2 years in scleroderma lung disease. Am J Respir Crit Care Med. 2007 Nov 15;176(10):1026-34. doi: 10.1164/rccm.200702-326OC. Epub 2007 Aug 23. PMID 17717203
- [Result] Strange C, Bolster MB, Roth MD, Silver RM, Theodore A, Goldin J, Clements P, Chung J, Elashoff RM, Suh R, Smith EA, Furst DE, Tashkin DP; Scleroderma Lung Study Research Group. Bronchoalveolar lavage and response to cyclophosphamide in scleroderma interstitial lung disease. Am J Respir Crit Care Med. 2008 Jan 1;177(1):91-8. doi: 10.1164/rccm.200705-655OC. Epub 2007 Sep 27. PMID 17901414
- [Result] Goldin JG, Lynch DA, Strollo DC, Suh RD, Schraufnagel DE, Clements PJ, Elashoff RM, Furst DE, Vasunilashorn S, McNitt-Gray MF, Brown MS, Roth MD, Tashkin DP; Scleroderma Lung Study Research Group. High-resolution CT scan findings in patients with symptomatic scleroderma-related interstitial lung disease. Chest. 2008 Aug;134(2):358-367. doi: 10.1378/chest.07-2444. Epub 2008 Jul 18. PMID 18641099
- [Result] Khanna D, Tseng CH, Furst DE, Clements PJ, Elashoff R, Roth M, Elashoff D, Tashkin DP; for Scleroderma Lung Study Investigators. Minimally important differences in the Mahler's Transition Dyspnoea Index in a large randomized controlled trial--results from the Scleroderma Lung Study. Rheumatology (Oxford). 2009 Dec;48(12):1537-40. doi: 10.1093/rheumatology/kep284. Epub 2009 Sep 23. PMID 19776222
- [Result] Goldin J, Elashoff R, Kim HJ, Yan X, Lynch D, Strollo D, Roth MD, Clements P, Furst DE, Khanna D, Vasunilashorn S, Li G, Tashkin DP. Treatment of scleroderma-interstitial lung disease with cyclophosphamide is associated with less progressive fibrosis on serial thoracic high-resolution CT scan than placebo: findings from the scleroderma lung study. Chest. 2009 Nov;136(5):1333-1340. doi: 10.1378/chest.09-0108. PMID 19892673
- [Result] Au K, Mayes MD, Maranian P, Clements PJ, Khanna D, Steen VD, Tashkin D, Roth MD, Elashoff R, Furst DE. Course of dermal ulcers and musculoskeletal involvement in systemic sclerosis patients in the scleroderma lung study. Arthritis Care Res (Hoboken). 2010 Dec;62(12):1772-8. doi: 10.1002/acr.20320. PMID 20740615
- [Derived] Volkmann ER, Wilhalme H, Good S, Kim GHJ, Goldin J, Roth MD, Tashkin DP. A composite endpoint for systemic sclerosis-associated interstitial lung disease: association with mortality in two clinical trial cohorts. Respir Res. 2025 Nov 28;26(1):337. doi: 10.1186/s12931-025-03401-8. PMID 41316297
- [Derived] Assassi S, Li N, Volkmann ER, Mayes MD, Runger D, Ying J, Roth MD, Hinchcliff M, Khanna D, Frech T, Clements PJ, Furst DE, Goldin J, Bernstein EJ, Castelino FV, Domsic RT, Gordon JK, Hant FN, Shah AA, Shanmugam VK, Steen VD, Elashoff RM, Tashkin DP. Predictive Significance of Serum Interferon-Inducible Protein Score for Response to Treatment in Systemic Sclerosis-Related Interstitial Lung Disease. Arthritis Rheumatol. 2021 Jun;73(6):1005-1013. doi: 10.1002/art.41627. Epub 2021 Apr 20. PMID 33350170
- [Derived] Kim GHJ, Tashkin DP, Lo P, Brown MS, Volkmann ER, Gjertson DW, Khanna D, Elashoff RM, Tseng CH, Roth MD, Goldin JG. Using Transitional Changes on High-Resolution Computed Tomography to Monitor the Impact of Cyclophosphamide or Mycophenolate Mofetil on Systemic Sclerosis-Related Interstitial Lung Disease. Arthritis Rheumatol. 2020 Feb;72(2):316-325. doi: 10.1002/art.41085. Epub 2019 Dec 26. PMID 31430058
- [Derived] Khanna D, Clements PJ, Volkmann ER, Wilhalme H, Tseng CH, Furst DE, Roth MD, Distler O, Tashkin DP. Minimal Clinically Important Differences for the Modified Rodnan Skin Score: Results from the Scleroderma Lung Studies (SLS-I and SLS-II). Arthritis Res Ther. 2019 Jan 16;21(1):23. doi: 10.1186/s13075-019-1809-y. PMID 30651141
- [Derived] Kafaja S, Clements PJ, Wilhalme H, Tseng CH, Furst DE, Kim GH, Goldin J, Volkmann ER, Roth MD, Tashkin DP, Khanna D. Reliability and minimal clinically important differences of forced vital capacity: Results from the Scleroderma Lung Studies (SLS-I and SLS-II). Am J Respir Crit Care Med. 2018 Mar 1;197(5):644-652. doi: 10.1164/rccm.201709-1845OC. Epub 2017 Nov 3. PMID 29099620
- [Derived] Namas R, Tashkin DP, Furst DE, Wilhalme H, Tseng CH, Roth MD, Kafaja S, Volkmann E, Clements PJ, Khanna D; Participants in the Scleroderma Lung Study I and members of the Scleroderma Lung Study II Research Group. Efficacy of Mycophenolate Mofetil and Oral Cyclophosphamide on Skin Thickness: Post Hoc Analyses From Two Randomized Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2018 Mar;70(3):439-444. doi: 10.1002/acr.23282. Epub 2018 Feb 9. PMID 28544580
- [Derived] Volkmann ER, Tashkin DP, Roth MD, Clements PJ, Khanna D, Furst DE, Mayes M, Charles J, Tseng CH, Elashoff RM, Assassi S. Changes in plasma CXCL4 levels are associated with improvements in lung function in patients receiving immunosuppressive therapy for systemic sclerosis-related interstitial lung disease. Arthritis Res Ther. 2016 Dec 30;18(1):305. doi: 10.1186/s13075-016-1203-y. PMID 28038680
- [Derived] Tashkin DP, Volkmann ER, Tseng CH, Roth MD, Khanna D, Furst DE, Clements PJ, Theodore A, Kafaja S, Kim GH, Goldin J, Ariolla E, Elashoff RM. Improved Cough and Cough-Specific Quality of Life in Patients Treated for Scleroderma-Related Interstitial Lung Disease: Results of Scleroderma Lung Study II. Chest. 2017 Apr;151(4):813-820. doi: 10.1016/j.chest.2016.11.052. Epub 2016 Dec 22. PMID 28012804
- [Derived] Tashkin DP, Roth MD, Clements PJ, Furst DE, Khanna D, Kleerup EC, Goldin J, Arriola E, Volkmann ER, Kafaja S, Silver R, Steen V, Strange C, Wise R, Wigley F, Mayes M, Riley DJ, Hussain S, Assassi S, Hsu VM, Patel B, Phillips K, Martinez F, Golden J, Connolly MK, Varga J, Dematte J, Hinchcliff ME, Fischer A, Swigris J, Meehan R, Theodore A, Simms R, Volkov S, Schraufnagel DE, Scholand MB, Frech T, Molitor JA, Highland K, Read CA, Fritzler MJ, Kim GHJ, Tseng CH, Elashoff RM; Sclerodema Lung Study II Investigators. Mycophenolate mofetil versus oral cyclophosphamide in scleroderma-related interstitial lung disease (SLS II): a randomised controlled, double-blind, parallel group trial. Lancet Respir Med. 2016 Sep;4(9):708-719. doi: 10.1016/S2213-2600(16)30152-7. Epub 2016 Jul 25. PMID 27469583
- [Derived] Tashkin DP, Volkmann ER, Tseng CH, Kim HJ, Goldin J, Clements P, Furst D, Khanna D, Kleerup E, Roth MD, Elashoff R. Relationship between quantitative radiographic assessments of interstitial lung disease and physiological and clinical features of systemic sclerosis. Ann Rheum Dis. 2016 Feb;75(2):374-81. doi: 10.1136/annrheumdis-2014-206076. Epub 2014 Dec 1. PMID 25452309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out between September 28, 2009, and January 14, 2013, at 14 University Medical Centers within the United States.
Groups:
- Mycophenolate Arm: Participants treated with oral mycophenolate mofetil for 2 years.
  Mycophenolate mofetil: 24 months of oral mycophenolate mofetil, up to a maximal dose of 1.5 grams twice daily as tolerated
- Cyclophosphamide Arm: Participants treated with oral cyclophosphamide for 1 year, followed by placebo for 1 year.
  Cyclophosphamide: 12 months of oral cyclophosphamide, up to a maximal dose of 2 mg/kg daily as tolerated
  Placebo: 12 months of placebo will be delivered to participants in the Cyclophosphamide arm during the second year in order to maintain the blind with the Mycophenolate arm, which receives drug for the entire 2 years.
Period: Overall Study
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Started | 69 | 73
Completed | 49 (53 subjects provided a 24 month outcome, 4 of whom had prematurely withdrawn from drug treatment.) | 37 (53 subjects provided a 24 month outcome, 16 of whom had prematurely withdrawn from drug treatment.)
Not Completed | 20 | 36
Not completed — Adverse Event | 7 | 15
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Non-compliance | 3 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 2
Not completed — Defined Treatment Failure | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm | Total
Number analyzed (Participants) | 69 | 73 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.7) | 52.0 (9.8) | 52.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 57 | 105
  Male | 21 | 16 | 37
Duration of scleroderma [Mean (Standard Deviation); unit: years] — Population: Only participants with available data included
  years
    number analyzed (Participants) | 67 | 72 | 139
    (all) | 2.6 (1.7) | 2.5 (1.8) | 2.6 (1.8)
Limited cutaneous scleroderma [Count of Participants; unit: Participants] | 26 | 33 | 59
Diffuse cutaneous scleroderma [Count of Participants; unit: Participants] | 43 | 40 | 83
modified-Rodnan Skin Score [Mean (Standard Deviation); unit: Score] — Skin score may range 0-51, with higher scores indicating more severe thickening
  Score | 15.3 (10.4) | 14.0 (10.6) | 14.7 (10.5)
FVC %-predicted [Mean (Standard Deviation); unit: Percent of predicted normal value] | 66.5 (9.1) | 66.5 (8.3) | 66.5 (9.9)
FEV1/FVC %-predicted [Mean (Standard Deviation); unit: Percent of predicted normal value] | 81.0 (5.5) | 83.3 (5.6) | 82.6 (5.6)
Total Lung Capacity [Mean (Standard Deviation); unit: Percent of predicted normal value] | 66.3 (10.0) | 65.5 (12.0) | 65.8 (11.1)
Single-Breath Diffusing Capacity [Mean (Standard Deviation); unit: Percent of predicted normal value] | 60.9 (11.8) | 61.0 (13.7) | 60.9 (12.8)
Mahler Dyspnea Index, mean focal score [Mean (Standard Deviation); unit: Score] — Scores range 0-12, with lower scores indicating worse dyspnea Population: Only participants with available data included
  Score
    number analyzed (Participants) | 65 | 68 | 133
    (all) | 7.3 (2.1) | 7.1 (2.3) | 7.2 (2.2)
SF-36 Physical component [Mean (Standard Deviation); unit: Score] — Score range 0-100, with lower scores indicating worse health status
  Score | 36.0 (10.0) | 35.6 (9.8) | 35.8 (9.9)
SF-36 Mental component [Mean (Standard Deviation); unit: Score] — Score range 0-100, with lower scores indicating worse health status
  Score | 49.1 (7.9) | 49.8 (10.0) | 49.4 (9.0)
HAQ disability index [Mean (Standard Deviation); unit: Score] — Score range 0-3, with higher scores indicating greater disability
  Score | 0.7 (0.6) | 0.7 (0.7) | 0.7 (0.7)
Quantitative extent of lung fibrosis on HRCT, for whole lung [Mean (Standard Deviation); unit: Score] — Score range 0 to 100, with higher score indicating greater lung involvement Population: Only participants with available data included
  Score
    number analyzed (Participants) | 66 | 71 | 137
    (all) | 8.3 (6.9) | 8.9 (7.0) | 8.6 (6.9)
Quantitative extent of lung fibrosis on HRCT, for lobe of maximum involvement [Mean (Standard Deviation); unit: Score] — Score range 0 to 100, with higher score indicating greater lung involvement Population: Only participants with available data included
  Score
    number analyzed (Participants) | 66 | 71 | 137
    (all) | 23.0 (20.2) | 22.6 (19.3) | 22.8 (19.6)
Quantitative extent of total insterstitial lung disease on HRCT, for whole lung [Mean (Standard Deviation); unit: Score] — Score range 0 to 100, with higher score indicating greater lung involvement Population: Only participants with available data included
  Score
    number analyzed (Participants) | 66 | 71 | 137
    (all) | 27.2 (13.2) | 31.6 (14.4) | 29.5 (14.0)
Quantitative extent of total insterstitial lung disease on HRCT, for lobe of maximum involvement [Mean (Standard Deviation); unit: Score] — Score range 0 to 100, with higher score indicating greater lung involvement Population: Only participants with available data included
  Score
    number analyzed (Participants) | 66 | 71 | 137
    (all) | 50.0 (20.9) | 52.3 (19.9) | 51.2 (20.3)
ANA(+) [Count of Participants; unit: Participants] — Population: Only participants with available data included
  Participants
    number analyzed (Participants) | 63 | 71 | 134
    (all) | 61 | 66 | 127
Topoisomerase-1(+) [Count of Participants; unit: Participants] — Population: Only participants with available data included
  Participants
    number analyzed (Participants) | 63 | 71 | 134
    (all) | 29 | 32 | 61
RNA Polymerase(+) [Count of Participants; unit: Participants] — Population: Only participants with available data included
  Participants
    number analyzed (Participants) | 63 | 71 | 134
    (all) | 9 | 9 | 18
Centromere(+) [Count of Participants; unit: Participants] — Population: Only participants with available data included
  Participants
    number analyzed (Participants) | 63 | 71 | 134
    (all) | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC), as a Percent of the Age, Height, Gender, and Ethnicity Adjusted Predicted Value
Description: The primary outcome is the course over time from baseline to 24 months for the FVC %-predicted. The FVC %-predicted represents the adjusted volume of air (adjusted as a percentage of the expected normal valued based on the participant's age, height, gender and ethnicity) that can be forcibly exhaled from the lungs after taking the deepest breath possible. The FVC %-predicted is reduced in patients with interstitial lung disease and is used as a measure of lung involvement and disease severity.
Time Frame: Measured at study Baseline and Months 3, 6, 12, 15, 18, 21, and 24
Population: Randomized participants with an acceptable baseline HRCT study (a pre-specified covariate) and at least one outcome measure
Measure: Mean (95% Confidence Interval); unit: FVC %-pred
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
FVC %-pred
  Baseline | 66.52 [64.55 to 68.49] | 66.52 [64.22 to 68.82]
  Month 3 | 66.22 [64.08 to 69.42] | 67.03 [64.64 to 69.42]
  Month 6: number analyzed (Participants) | 60 | 56
  Month 6 | 68.02 [65.55 to 70.49] | 67.86 [65.27 to 70.45]
  Month 9: number analyzed (Participants) | 54 | 51
  Month 9 | 68.11 [65.55 to 70.67] | 69.42 [66.34 to 72.50]
  Month 12: number analyzed (Participants) | 59 | 51
  Month 12 | 68.43 [65.48 to 71.38] | 69.86 [66.82 to 72.90]
  Month 15: number analyzed (Participants) | 51 | 44
  Month 15 | 69.84 [67.14 to 72.54] | 71.94 [68.40 to 75.48]
  Month 18: number analyzed (Participants) | 49 | 46
  Month 18 | 70.57 [67.57 to 73.57] | 72.57 [69.53 to 75.61]
  Month 21: number analyzed (Participants) | 47 | 40
  Month 21 | 70.87 [67.91 to 73.83] | 72.55 [69.18 to 75.92]
  Month 24: number analyzed (Participants) | 53 | 51
  Month 24 | 69.65 [66.53 to 72.77] | 70.15 [66.88 to 73.42]
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in the FVC %-predicted. Covariates were %-predicted FVC, HRCT-defined extent of lung fibrosis in the lobe of maximum involvement, and terms for time-trend, treatment and treatment-time trend interactions; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 2: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; The inferential joint model, as described for the primary analysis, was used to estimate the change from baseline to 24 months for the FVC %-predicted for each treatment arm independently; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 3: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; Based on the absolute difference between the value of FVC %-predicted at baseline and at 24 months for each subject who returned for a 24-month assessment, a frequency distributions was prepared, stratified by treatment arm, to assess the relative distribution of subjects who either had improvements or worsening in the FVC %-predicted; Test type: Superiority or Other; p = 0.55, Fisher Exact — The threshold for statistical significance was a P-Value of </=0.05

2. Secondary Outcome: Total Lung Capacity (TLC), as a Percent of the Age, Height, Gender, and Ethnicity Adjusted Predicted Value
Description: The TLC represents the total volume of air within the lung after taking the deepest breath possible and the TLC %-predicted represents the TLC expressed as a percentage of the expected normal valued based on the participant's age, height, gender and ethnicity. The TLC %-predicted is reduced in patients with interstitial lung disease and is used as a measure of disease severity.
Time Frame: Measured at study entry and Months 6, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: TLC %-pred
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
TLC %-pred
  Baseline | 66.16 [63.74 to 68.58] | 65.49 [62.72 to 68.26]
  Month 6: number analyzed (Participants) | 60 | 56
  Month 6 | 67.84 [65.35 to 70.33] | 67.39 [64.30 to 70.48]
  Month 12: number analyzed (Participants) | 57 | 54
  Month 12 | 67.31 [64.45 to 70.17] | 68.25 [64.93 to 71.57]
  Month 18: number analyzed (Participants) | 49 | 46
  Month 18 | 68.50 [65.45 to 71.55] | 69.63 [65.65 to 73.61]
  Month 24: number analyzed (Participants) | 53 | 51
  Month 24 | 68.24 [64.99 to 71.49] | 66.97 [63.42 to 70.52]
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in the TLC %-predicted; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05

3. Secondary Outcome: Single-breath Diffusing Capacity for Carbon Monoxide (DLCO), as a Percent of the Age, Height, Gender, and Ethnicity Adjusted Predicted Value
Description: The DLCO is a pulmonary function test that measures the capacity for the lung to carry out gas exchange between the inhaled breath and the pulmonary capillary blood vessels and the DLCO %-predicted represents the DLCO expressed as a percentage of the expected normal valued based on the participant's age, height, gender and ethnicity. The DLCO %-predicted is reduced in patients with interstitial lung disease and is used as a measure of disease severity.
Time Frame: Measured at study entry and Months 3, 6, 12, 15, 18, 21, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: DLCO %-pred
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
DLCO %-pred
  Baseline | 53.99 [51.35 to 56.63] | 54.05 [50.80 to 57.30]
  Month 3: number analyzed (Participants) | 62 | 64
  Month 3 | 53.38 [50.48 to 56.28] | 51.92 [48.34 to 55.50]
  Month 6: number analyzed (Participants) | 60 | 56
  Month 6 | 54.86 [51.27 to 58.45] | 50.87 [46.84 to 56.28]
  Month 9: number analyzed (Participants) | 54 | 50
  Month 9 | 54.13 [50.50 to 57.76] | 51.55 [47.09 to 56.01]
  Month 12: number analyzed (Participants) | 58 | 51
  Month 12 | 55.32 [51.31 to 59.33] | 53.12 [48.38 to 57.86]
  Month 15: number analyzed (Participants) | 51 | 44
  Month 15 | 57.77 [54.20 to 61.34] | 53.62 [48.29 to 58.95]
  Month 18: number analyzed (Participants) | 49 | 44
  Month 18 | 56.62 [52.84 to 60.40] | 55.9 [50.82 to 60.98]
  Month 21: number analyzed (Participants) | 47 | 40
  Month 21 | 55.47 [51.39 to 59.55] | 54.26 [49.29 to 59.23]
  Month 24: number analyzed (Participants) | 52 | 48
  Month 24 | 55.31 [51.64 to 58.98] | 52.90 [48.71 to 57.09]
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in the DLCO %-predicted; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 2: Comparison: Mycophenolate Arm; The inferential joint model, as described for the primary analysis, was used to estimate the change from baseline to 24 months for the DLCO %-predicted for each treatment arm independently; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05

4. Secondary Outcome: Fibrosis Score, as Measured by Thoracic High Resolution Computerized Tomography (HRCT)
Description: Imaging of the whole lung (WL) is performed using a volumetric high resolution computerized tomography (HRCT) scan, which is then analyzed using a computer algorithm to determine the percentage of overall pixels exhibiting features characteristic for quantitative lung fibrosis (QLF). Higher percentages for QLF-WL therefore represent greater involvement by lung fibrosis.
Time Frame: Measured at baseline and Month 24
Population: Analysis was carried out in the subset of subjects that had measurable HRCT scans at both study entry and 24 months
Measure: Mean (95% Confidence Interval); unit: % of lung exhibiting QLF
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
% of lung exhibiting QLF
  Baseline: number analyzed (Participants) | 66 | 71
  Baseline | 8.25 [6.58 to 9.92] | 8.91 [7.26 to 10.56]
  Month 24: number analyzed (Participants) | 51 | 47
  Month 24 | 7.99 [6.14 to 9.84] | 8.48 [6.33 to 10.63]
Statistical Analysis 1: Comparison: Mycophenolate Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in the Quantitative Lung Fibrosis Score for the whole lung (QLF-WL); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05

5. Secondary Outcome: Transitional Dyspnea Index Score
Description: Change in breathlessness was assessed using the Transitional Dyspnea Index, which compares current symptoms to those at baseline. Total score ranges from - 9 to + 9. The lower the score, the more deterioration in severity of dyspnea.
Time Frame: Measured at Months 6, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Transitional Dyspnea Index Score
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
Transitional Dyspnea Index Score
  Month 6: number analyzed (Participants) | 52 | 50
  Month 6 | 0.74 [-0.07 to 1.55] | 0.31 [-0.43 to 1.05]
  Month 12: number analyzed (Participants) | 49 | 47
  Month 12 | 1.17 [0.23 to 2.11] | 1.23 [0.14 to 2.32]
  Month 18: number analyzed (Participants) | 42 | 35
  Month 18 | 0.91 [-0.01 to 1.83] | 1.78 [0.47 to 3.09]
  Month 24: number analyzed (Participants) | 40 | 39
  Month 24 | 1.86 [0.62 to 3.10] | 2.09 [0.80 to 3.38]
Statistical Analysis 1: Comparison: Mycophenolate Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in dyspnea as measured by the Transitional Dyspnea Index Score; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 2: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; The inferential joint model, as described for the primary analysis, was used to estimate the change from baseline to 24 months for dyspnea using the Transitional Dyspnea Index Score for each treatment arm independently; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05

6. Secondary Outcome: Health-related Quality of Life as Measured by the Patient Responses to the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI asks questions related to 8 activity domains (dressing, arising, eating, walking, hygiene, reach, grip, and common daily activities) with the patient's capacity to carry out each activity scored from 0 to 3. Scores across all domains are averaged and a higher score represents greater disability.
Time Frame: Measured at study entry and Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: The analysis population contains all of those with data available at the defined time point.
Measure: Mean (Standard Deviation); unit: HAQ-DI Total Score
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
HAQ-DI Total Score
  Baseline | 0.71 (0.62) | 0.74 (0.73)
  Month 3: number analyzed (Participants) | 66 | 65
  Month 3 | 0.83 (0.72) | 0.64 (0.67)
  Month 6: number analyzed (Participants) | 60 | 58
  Month 6 | 0.75 (0.71) | 0.58 (0.65)
  Month 9: number analyzed (Participants) | 54 | 55
  Month 9 | 0.66 (0.66) | 0.65 (0.62)
  Month 12: number analyzed (Participants) | 58 | 55
  Month 12 | 0.64 (0.67) | 0.56 (0.60)
  Month 15: number analyzed (Participants) | 51 | 45
  Month 15 | 0.58 (0.62) | 0.62 (0.63)
  Month 18: number analyzed (Participants) | 50 | 47
  Month 18 | 0.55 (0.55) | 0.55 (0.66)
  Month 21: number analyzed (Participants) | 49 | 40
  Month 21 | 0.65 (0.65) | 0.48 (0.53)
  Month 24: number analyzed (Participants) | 53 | 53
  Month 24 | 0.62 (0.69) | 0.57 (0.68)

7. Secondary Outcome: Skin Involvement, as Measured by the Modified Rodnam Skin Thickness Scores (mRSS)
Description: Skin thickness is quantified using the modified Rodnan measurement method (mRSS), with a scale that ranges from 0 (no skin involvement) to a maximum of 51. The reported skin score is determined by a clinical assessment of skin thickness, which is performed by a trained reader, and represents the sum of individual assessments that are made in each of 17 body areas. Each area is given a score in the range of 0-3 (0 = normal; 1= mild thickness; 2 = moderate; 3 = severe thickness). A higher score represents more severe skin involvement.
Time Frame: Measured at baseline and Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mRSS score
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
mRSS score
  Baseline | 15.32 [12.85 to 17.79] | 14.04 [11.58 to 16.50]
  Month 3: number analyzed (Participants) | 65 | 65
  Month 3 | 16.03 [13.44 to 18.62] | 12.85 [10.17 to 15.53]
  Month 6: number analyzed (Participants) | 60 | 58
  Month 6 | 14.37 [11.75 to 16.99] | 11.95 [9.27 to 14.63]
  Month 9: number analyzed (Participants) | 54 | 54
  Month 9 | 14.33 [11.62 to 17.04] | 10.61 [8.27 to 12.95]
  Month 12: number analyzed (Participants) | 58 | 55
  Month 12 | 12.45 [10.05 to 14.85] | 9.47 [7.35 to 11.59]
  Month 15: number analyzed (Participants) | 51 | 45
  Month 15 | 12.43 [10.08 to 14.78] | 9.80 [7.66 to 11.94]
  Month 18: number analyzed (Participants) | 50 | 47
  Month 18 | 11.98 [9.48 to 14.48] | 9.87 [7.60 to 12.14]
  Month 21: number analyzed (Participants) | 49 | 40
  Month 21 | 11.22 [8.74 to 13.70] | 8.50 [6.19 to 10.81]
  Month 24: number analyzed (Participants) | 53 | 53
  Month 24 | 11.40 [8.91 to 13.89] | 7.87 [5.85 to 9.89]
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; A modified intention-to-treat inferential joint model combined a mixed-effects model for longitudinal outcomes and a survival model to handle non-ignorable missing data due to study dropout, treatment failure, or death, to assess the course over time, from baseline to 24 months, for the change in modified Rodnan Skin Score (mRSS); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 2: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; The inferential joint model, as described for the primary analysis, was used to estimate the change from baseline to 24 months for the modified Rodnan Skin Score for each treatment arm independently; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was a P-Value of </=0.05
Statistical Analysis 3: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; Based on the absolute difference between the value of the mRSS at baseline and at 24 months for each subject who returned for a 24-month assessment, a frequency distributions was prepared, stratified by treatment arm, to assess the relative distribution of subjects who either had improvements or worsening in the mRSS; Test type: Superiority or Other; p > 0.05, Fisher Exact — The threshold for statistical significance was a P-Value of </=0.05

8. Secondary Outcome: Toxicity, as Measured by Adverse Events, Serious Adverse Events, and Death
Time Frame: Measured throughout the 2-year study
Measure: Count of Participants; unit: Participants
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
Participants
  Leukopenia (<2.5x10^3 WBC/microliter) | 4 | 30
  Neutropenia (<1.0x10^3 neutrophils/microliter) | 3 | 7
  Anemia (Hgb <10 g/dl) | 8 | 13
  Thrombocytopenia (<100x10^3 platelets/microliter) | 0 | 4
  Hematuria (>10 RBC/high power field) | 3 | 2
  Pneumonia | 5 | 4
  SAE-Total | 27 | 22
  SAE-related to treatment | 3 | 7
  Deaths | 5 | 11
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; Fisher's Exact Test was utilized to compare the number of participants with a protocol-defined adverse event of interest, SAE or death between the MMF and CYC treatment arms; Test type: Superiority or Other; p < 0.05, Fisher Exact — The threshold for statistical significance was a P-Value of </=0.05; The threshold for statistical significance was met only for the frequency of leukopenia and thrombocytopenia, but not for total SAE or death

9. Secondary Outcome: Tolerability, as Assessed by the Time to Withdrawal From the Study Drug or Meeting Protocol-defined Criteria for Treatment Failure.
Description: The number of participants who remained in the study at the listed time points are reported
Time Frame: Continuous assessment from randomization to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Number analyzed (Participants) | 69 | 73
Participants
  Baseline | 69 | 73
  Month 3 | 66 | 64
  Month 6 | 58 | 56
  Month 9 | 55 | 51
  Month 12 | 52 | 46
  Month 15 | 52 | 44
  Month 18 | 49 | 42
  Month 21 | 49 | 39
  Month 24 | 49 | 38
Statistical Analysis 1: Comparison: Mycophenolate Arm vs Cyclophosphamide Arm; A log-rank test was utilized to assess differences between the MMF and CYC treatment arms with respect to the time to withdrawal from study drug or meeting protocol-defined criteria for treatment failure; Test type: Superiority or Other; p = 0.019, Log Rank — The threshold for statistical significance was a P-Value of </=0.05

ADVERSE EVENTS:
Time Frame: Randomization to withdrawal from taking study drug or completion of the 24 month treatment protocol.
Description: An organ system designation was developed for the study and applied in a systematic manner to all adverse event assessments
Arm/Group | Mycophenolate Arm | Cyclophosphamide Arm
Serious Adverse Events (participants affected / at risk) | 27/69 | 22/73
Other Adverse Events (participants affected / at risk) | 68/69 | 71/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Arm (N=69) | Cyclophosphamide Arm (N=73)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal and Bladder (Renal and urinary disorders) | 1 | 1
Syncope and Seizure (Nervous system disorders) | 2 | 0
Hematologic (Blood and lymphatic system disorders) | 1 | 2
Gastrointestinal (Gastrointestinal disorders) | 2 | 4
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 | 3
Respiratory Infection (Infections and infestations) | 2 | 7
Respiratory Events (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Cardiac (Cardiac disorders) | 8 | 8
Weakness (General disorders) | 0 | 1
Medication Reaction (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Elective Surgery (Surgical and medical procedures) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Arm (N=69) | Cyclophosphamide Arm (N=73)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Immune disorder (Immune system disorders) | 2 | 4
Vision and hearing (Ear and labyrinth disorders) | 2 | 6
Hepatobiliary (Hepatobiliary disorders) | 6 | 4
Procedures (Surgical and medical procedures) | 6 | 5
Psychiatric (Psychiatric disorders) | 10 | 9
Injury, Poisoning and Procedural (Injury, poisoning and procedural complications) | 8 | 10
Nervous System (Nervous system disorders) | 12 | 9
Reproductive and Breast (Reproductive system and breast disorders) | 15 | 12
Metabolism and Nutrition (Metabolism and nutrition disorders) | 11 | 22
Vascular (Vascular disorders) | 19 | 22
Cardiac (Cardiac disorders) | 18 | 21
Renal and Urinary (Renal and urinary disorders) | 26 | 27
General (General disorders) | 31 | 33
Skin and Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 35 | 43
Musculoskeletal and Connective Tissue (Musculoskeletal and connective tissue disorders) | 34 | 34
Blood and Lymphatic (Blood and lymphatic system disorders) | 20 | 47
Respiratory and Thoracic (Respiratory, thoracic and mediastinal disorders) | 46 | 45
Gastrointestinal (Gastrointestinal disorders) | 47 | 40
Infections and Infestations (Infections and infestations) | 52 | 57

LIMITATIONS AND CAVEATS:
While the rate of premature withdrawal from taking study drug was significant, this was anticipated in the study design and addressed by the sample size and the use of the mixed model statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No